CLINICAL TRIAL: NCT04249440
Title: Preoperative Systemic Therapy Versus Upfront Surgery in HER2 Positive Early Breast Cancer: a Prospective Nested Case-control Study in Real World
Brief Title: Preoperative Systemic Therapy vs Upfront Surgery in HER2 Positive Early Breast Cancer
Status: Completed | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, YU Xingfei, Department of Breast Tumor Surgery, Zhejiang Cancer Hospital
Other Study IDs: HER2-RWSNeo
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; HER2; Preoperative Systemic Treatment
Keywords: breast cancer; HER2; preoperative systemic treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PST: patient accepts preoperative systemic treatment as upfront strategy
  Interventions: Procedure: Preoperative systemic treatment
- upfront surgery: patient accepts upfront surgery and run postoperative systemic treatment

INTERVENTIONS:
Procedure: Preoperative systemic treatment — neoadjuvant chemotherapy combined with trastuzumab as preoperative systemic treatment
  Other Names: neoadjuvant treatment
  Groups: PST

SUMMARY:
Preoperative systemic treatment can make patients getting more opportunity for breast-conserving surgery, down-staging and new drugs developing. It is particularly common in human epidermal growth factor receptor 2 (HER2)-over expressing subtype for as high as 40%~60% pCR rate of such a population. Even though, in NSABP B18/27 trials, it had been proved that PST could not improve either disease-free survival (DFS) or overall survival (OS) comparing with postoperatively systemic treatment in total population. We designed a real-world study to investigate the prognosis of anti-HER2 treatment combined with chemotherapy preoperatively versus postoperatively in HER2-positive early breast cancer

DETAILED DESCRIPTION:
Patients with a diagnosis of HER2 positive early invasive breast cancer (cT1-3N0-1M0), from January 2012 to December 2014 were identified and enrolled continuously. The conditions of HER2-positive expression of primary breast cancer were defined as follows: HER2 3+ by immunohistochemical (IHC) method or HER2 2+ by IHC with a further positive result by fluorescence in situ hybridization (FISH). According to the real upfront treatment, all eligible patients were classified as PST group and surgery group. All the patients accepted standard one-year trastuzumab as anti-HER2 treatment combined with chemotherapy. In the PST group, the effect was evaluated according to RECIST1.1 every two cycles, the patients with clinical complete response (cCR) or partial response (PR) would receive the whole course of chemotherapy, those with stable disease (SD) or progressive disease (PD) would receive surgery promptly. After surgery, all patients underwent irradiation and endocrine therapies if necessary. The pCR was defined as the absence of infiltrating residual invasive disease in the breast and axillary nodes. For those non-pCR patients after PST, intensive adjuvant chemotherapy was not routine treatment except patients with progressive disease.The primary endpoint was DFS defined as the time from enrollment to local, regional, or distant recurrences; the occurrence of contralateral breast cancer; or death without evidence of breast cancer. Patients suffered disease progress becoming inoperable before surgery were counted as local treatment failures. The second endpoint was OS defined as the time from study entry to death from any cause. All the endpoints were compared between PST group and upfront surgery group, also further analysis according to pathological response status stratified in PST group.

ELIGIBILITY:
Inclusion Criteria:

1. HER2 positive
2. early invasive breast cancer (cT1-3N0-1M0)
3. using one-year trastuzumab as anti-HER2 treatment

Exclusion Criteria:

1. Exclude metastasis and recurrent breast cancer
2. using trastuzumab less than a year

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2 positive early invasive breast cancer, using trastuzumab for one year both in neoadjuvant or adjuvant setting.
Sampling Method: Non-Probability Sample
Enrollment: 1067 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 5 years
  as the time from enrollment to local, regional, or distant recurrences; the occurrence of contralateral breast cancer; or death without evidence of breast cancer

SECONDARY OUTCOMES:
Overall survival | 5 years
  the time from study entry to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Xingfei Yu, M.D., Principal Investigator — Zhejiang Cancer Hospital

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to others

REFERENCES:
- [Derived] Yu X, Wang C, Zheng Y, Miao B, Hu J, Shao X, Sheng L, Lin J, Ding Y, Xuan H, Ding Y, Gong L, Feng W, Qin C, Chen D, Yu Y, Yang H. Preoperative Systemic Therapy Versus Upfront Surgery in HER2-Positive Breast Cancer in the Real World. Front Oncol. 2021 Jul 28;11:704842. doi: 10.3389/fonc.2021.704842. eCollection 2021. PMID 34395277